CLINICAL TRIAL: NCT02596191
Title: Tools for Therapeutic Evaluation in Charcot-Marie-Tooth Disease Type 1A: Outcome Measures and Biomarkers
Acronym: CMT-TOOLS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2014-10
Record Dates: First submitted 2015-10-30; First posted 2015-11-04 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Charcot-Marie-Tooth Disease Type 1A
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- patients with mild CMT 1A disease (Experimental): Charcot-Marie-Tooth Neuropathy Score between 1 and 10
  Interventions: Other: Clinical evaluation; Other: electrophysiological record; Other: Muscle MRI; Other: blood samples analysis
- patients with moderate CMT 1A disease (Experimental): Charcot-Marie-Tooth Neuropathy Score between 11 and 20
  Interventions: Other: Clinical evaluation; Other: electrophysiological record; Other: Muscle MRI; Other: blood samples analysis
- patients with severe CMT 1A disease (Experimental): Charcot-Marie-Tooth Neuropathy Score ≥21
  Interventions: Other: Clinical evaluation; Other: electrophysiological record; Other: Muscle MRI; Other: blood samples analysis
- control group (Other): Healthy volunteers
  Interventions: Other: Muscle MRI; Other: blood samples analysis

INTERVENTIONS:
Other: Clinical evaluation
  Arms: patients with mild CMT 1A disease; patients with moderate CMT 1A disease; patients with severe CMT 1A disease
Other: electrophysiological record
  Arms: patients with mild CMT 1A disease; patients with moderate CMT 1A disease; patients with severe CMT 1A disease
Other: Muscle MRI
Other: blood samples analysis

SUMMARY:
This is a 2-year follow-up study of a cohort of 60 CMT1A patients. The objective is to identify markers allowing to better understand the phenotypic variability observed on patients with CMT1A, to identify predictive markers of the disease's progression and to provide validated measurement tools that can be used as outcome measures in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CMT 1A disease
* Diagnosis of CMT 1A confirmed by genotyping (duplication of the 17p11.2 region)

Exclusion Criteria:

* Patients suffering from co-morbidity at the origin of peripheral neuropathy (diabetes, hypothyroidism, renal insufficiency, drugs...) or muscle, articular, rheumatological disease
* With HIV or cancer
* With a significant progressive disease in the previous month
* With a contra-indication for MRI
* With a dislocation, fracture, or recent surgery (less than 6 months before inclusion)
* with alcohol or psychoactive substances abuse
* Treated by an anti-inflammatory drug over the past four weeks
* Pregnant or breastfeeding women
* Homeless patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06-06 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2027-12-05 (Estimated)

PRIMARY OUTCOMES:
Change of functional scores | 3 months, 12 months and 24 months
  several functional scores to evaluate the severity and the progression of the disease will be performed and compared (CMTNDS)
Change of functional scores | 3 months, 12 months and 24 months
  several functional scores to evaluate the severity and the progression of the disease will be performed and compared (CMTNS)
Change of functional scores | 3 months, 12 months and 24 months
  several functional scores to evaluate the severity and the progression of the disease will be performed and compared (CMTNS2)
Change of functional scores at | 3 months, 12 months and 24 months
  several functional scores to evaluate the severity and the progression of the disease will be performed and compared (ONLS)

SECONDARY OUTCOMES:
Walkin test | 12 months and 24 months
  Use of connected soles for walking test (Digitsole)

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (2):
- France (2):
  - Assistance Publique Hôpitaux de Marseille, Marseille
  - CHU Gui de Chauliac, CHU MONTPELLIER, Montpellier